CLINICAL TRIAL: NCT01318499
Title: Clinical Evaluation of Nepafenac Ophthalmic Suspension, 0.3% Compared to Nepafenac Ophthalmic Suspension 0.1% and Vehicle for Prevention and Treatment of Ocular Inflammation and Pain Associated With Cataract Surgery
Brief Title: Nepafenac 0.3% Two Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-11-003
Record Dates: First submitted 2011-03-15; First posted 2011-03-18 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Cataract
Keywords: cataract; inflammation; pain; inflammatory cells; aqueous flare
MeSH Terms: conditions — Cataract; Inflammation; Pain | interventions — nepafenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nepafenac 0.3% (Experimental): Nepafenac Ophthalmic Suspension, 0.3%, one drop in affected eye once daily, for 16 days, beginning one day prior to surgery, continuing on the day of surgery, and for 14 days following surgery. An additional drop was administered between 30-120 minutes prior to surgery.
  Interventions: Drug: Nepafenac Ophthalmic Suspension, 0.3%
- Nepafenac 0.1% (Active Comparator): Nepafenac Ophthalmic Suspension, 0.1%, one drop in affected eye once daily, for 16 days, beginning one day prior to surgery, continuing on the day of surgery, and for 14 days following surgery. An additional drop was administered between 30-120 minutes prior to surgery.
  Interventions: Drug: Nepafenac Ophthalmic Suspension, 0.1%
- Nepafenac Vehicle 0.3% (Placebo Comparator): Nepafenac Vehicle 0.3%, one drop in affected eye once daily, for 16 days, beginning one day prior to surgery, continuing on the day of surgery, and for 14 days following surgery. An additional drop was administered between 30-120 minutes prior to surgery.
  Interventions: Other: Nepafenac Vehicle 0.3%

INTERVENTIONS:
Drug: Nepafenac Ophthalmic Suspension, 0.3% — Nepafenac Ophthalmic Suspension, 0.3%, one drop in affected eye once daily, for 16 days. An additional drop was administered between 30-120 minutes prior to surgery.
  Arms: Nepafenac 0.3%
Drug: Nepafenac Ophthalmic Suspension, 0.1% — Nepafenac Ophthalmic Suspension, 0.1%, one drop in affected eye once daily, for 16 days. An additional drop was administered between 30-120 minutes prior to surgery.
  Other Names: NEVANAC®
  Arms: Nepafenac 0.1%
Other: Nepafenac Vehicle 0.3% — Nepafenac Vehicle 0.3%, one drop in affected eye once daily, for 16 days. An additional drop was administered between 30-120 minutes prior to surgery.
  Arms: Nepafenac Vehicle 0.3%

SUMMARY:
The purpose of this study was to assess the safety and efficacy of Nepafenac Ophthalmic Suspension, 0.3% for the prevention and treatment of inflammation (swelling and redness) and pain in the eye after cataract extraction.

ELIGIBILITY:
Inclusion Criteria:

* Planned cataract extraction by phacoemulsification with the implantation of a posterior chamber intraocular lens;
* Patients who, in the opinion of the Investigator, would have improvement in best-corrected visual acuity after surgery;
* Able to understand and sign an informed consent;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Use of topical ocular, inhaled or systemic nonsteroidal anti-inflammatory drugs within 7 days of surgery, with the exception of the allowed low dose of aspirin (up to 100 mg) prior to surgery and through study exit;
* Use of topical ocular, inhaled or systemic steroids within 14 days prior to surgery and through study exit;
* History of chronic or recurrent inflammatory eye disease (eg, iritis, scleritis, uveitis, iridocyclitis, rubeosis iridis) in the operative eye;
* Diabetic retinopathy in the operative eye;
* Known or suspected allergy or hypersensitivity to non-steroidal anti-inflammatory drugs (NSAIDs), or to any component of the test article;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1342 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized from 37 investigational sites in the US.
Pre-assignment Details: Of the 1342 enrolled patients, 60 withdrew before the start of dosing. Baseline characteristics are presented on all randomized patients with at least one postoperative assessment (intent-to-treat): 1257
Period: Overall Study
Arm/Group | Nepafenac 0.3% | Nepafenac 0.1% | Nepafenac Vehicle 0.3%
Started | 540 | 534 | 268
Completed | 475 | 458 | 121
Not Completed | 65 | 76 | 147
Not completed — Adverse Event | 16 | 11 | 6
Not completed — Pt Decision Unrelated to Adverse Event | 1 | 1 | 2
Not completed — Noncompliance | 2 | 3 | 0
Not completed — Treatment Failure | 19 | 19 | 101
Not completed — Protocol Violation | 2 | 4 | 2
Not completed — Patient Did Not Use Study Medication | 18 | 28 | 14
Not completed — Other | 7 | 10 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepafenac 0.3% | Nepafenac 0.1% | Nepafenac Vehicle 0.3% | Total
Number analyzed (Participants) | 512 | 493 | 252 | 1257
Age Continuous [Mean (Standard Deviation); unit: years] | 69.3 (9.26) | 69.4 (9.15) | 69.3 (9.6) | 69.3 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 301 | 142 | 725
  Male | 230 | 192 | 110 | 532
Region of Enrollment [Number; unit: participants]
  United States | 512 | 493 | 252 | 1257

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Cured at Day 14, Nepafenac 0.3% vs. Nepafenac Vehicle 0.3%
Description: Ocular inflammation was assessed by the investigator during slit lamp examination. Aqueous cells were scored on a 5-unit scale from 0 (none) to 4 (> 30 cells), and aqueous flare (protein escaping from dilated vessels) was scored on a 4-unit scale from 0 (no visible flare when compared with the normal eye) to 3 (severe - very dense flare). To be considered cured, the patient must have had a score of 0 for both aqueous cells and aqueous flare.
Time Frame: Day 14 postoperative
Population: All randomized patients with at least one postoperative assessment (intent-to-treat), last observation carried forward.
Measure: Number; unit: Percentage of patients
Arm/Group | Nepafenac 0.3% | Nepafenac Vehicle 0.3%
Number analyzed (Participants) | 512 | 252
Percentage of patients | 64.6 | 25.0

2. Secondary Outcome: Percentage of Patients Cured at Day 7, Nepafenac 0.3% vs. Nepafenac 0.1%
Description: as for outcome 1
Time Frame: Day 7 postoperative
Population: All randomized patients with at least one postoperative assessment (intent-to-treat), last observation carried forward.
Measure: Number; unit: Percentage of patients
Arm/Group | Nepafenac 0.3% | Nepafenac 0.1%
Number analyzed (Participants) | 512 | 493
Percentage of patients | 31.3 | 30.8

3. Post Hoc Outcome: Cumulative Percent Clinical Success by Visit
Description: Ocular inflammation was assessed by the investigator during slit lamp examination. Aqueous cells were scored on a 5-unit scale from 0 (none) to 4 (> 30 cells), and aqueous flare (protein escaping from dilated vessels) was scored on a 4-unit scale from 0 (no visible flare when compared with the normal eye) to 3 (severe - very dense flare). Clinical success occurred when the cell grade was ≤ 1 (0-5 cells) and flare grade was = 0. To be included in the cumulative summary at a visit, a patient must have been declared a clinical success at the visit and remained a clinical success at all subsequent visits.
Time Frame: Day 1, Day 3, Day 7, Day 14
Population: All randomized patients with at least one post-operative assessment (intent-to-treat).
Measure: Number; unit: Percentage of patients
Arm/Group | Nepafenac 0.3% | Nepafenac 0.1% | Nepafenac Vehicle 0.3%
Number analyzed (Participants) | 512 | 493 | 252
Percentage of patients
  Day 1 | 18.9 | 15.0 | 12.3
  Day 3 | 43.9 | 35.9 | 18.7
  Day 7 | 71.9 | 62.5 | 29.4
  Day 14 | 84.8 | 81.3 | 37.7

4. Other Pre Specified Outcome: Cumulative Percentage of Patients Cured by Visit
Description: Ocular inflammation was assessed by the investigator during slit lamp examination. Aqueous cells were scored on a 5-unit scale from 0 (none) to 4 (> 30 cells), and aqueous flare (protein escaping from dilated vessels) was scored on a 4-unit scale from 0 (no visible flare when compared with the normal eye) to 3 (severe - very dense flare). To be considered cured, the patient must have had a score of 0 for both aqueous cells and aqueous flare. To be included in the cumulative summary at a visit, a patient must have been declared cured at the visit and remained cured at all subsequent visits.
Time Frame: Day 1, Day 3, Day 7, Day 14
Population: All randomized patients with at least one postoperative assessment (intent-to-treat), last observation carried forward.
Measure: Number; unit: Percentage of patients
Groups:
- Nepafenac 0.3% Vehicle: Nepafenac Vehicle 0.3%, one drop in affected eye once daily, for 16 days, beginning one day prior to surgery, continuing on the day of surgery, and for 14 days following surgery. An additional drop was administered between 30-120 minutes prior to surgery.
Arm/Group | Nepafenac 0.3% | Nepafenac 0.1% | Nepafenac 0.3% Vehicle
Number analyzed (Participants) | 512 | 493 | 252
Percentage of patients
  Day 1 | 0.4 | 1.8 | 0.4
  Day 3 | 6.4 | 7.1 | 3.2
  Day 7 | 31.3 | 30.8 | 10.3
  Day 14 | 64.6 | 65.3 | 25.0

5. Other Pre Specified Outcome: Cumulative Percentage of Patients Pain Free by Visit
Description: Ocular pain was assessed by the patient on a 6-unit scale from 0 (none; absence of positive sensation), to 5 (severe; intense ocular, periocular or radiating pain requiring prescription analgesic). Pain free was defined as an ocular pain assessment score of 0. To be included in the cumulative summary at a visit, a patient must have been declared pain free at the visit and remained pain free at all subsequent visits.
Time Frame: Day 1, Day 3, Day 7, Day 14
Population: All randomized patients with at least one postoperative assessment (intent-to-treat), last observation carried forward.
Measure: Number; unit: Percentage of patients
Arm/Group | Nepafenac 0.3% | Nepafenac 0.1% | Nepafenac 0.3% Vehicle
Number analyzed (Participants) | 512 | 493 | 252
Percentage of patients
  Day 1 | 65.2 | 61.9 | 17.5
  Day 3 | 77.3 | 75.9 | 25.8
  Day 7 | 84.8 | 83.0 | 31.7
  Day 14 | 89.1 | 89.0 | 40.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: The safety population includes all patients who received study medication, or potentially received study medication: 1282. At each study visit, the patient received an ocular exam, and any changes in ocular and systemic medications and/or systemic diseases/conditions since surgery were recorded.
Arm/Group | Nepafenac 0.3% | Nepafenac 0.1% | Nepafenac Vehicle 0.3%
Serious Adverse Events (participants affected / at risk) | 5/522 | 4/506 | 0/254
Other Adverse Events (participants affected / at risk) | 0/522 | 0/506 | 0/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nepafenac 0.3% (N=522) | Nepafenac 0.1% (N=506) | Nepafenac Vehicle 0.3% (N=254)
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 — Not related
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 — Not related
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Not related
Endophthalmitis (Infections and infestations) | 1 | 0 | 0 — Not related
Hypopyon (Infections and infestations) | 1 | 0 | 0 — Not related
Lens dislocation (Eye disorders) | 1 | 0 | 0 — Not related
Retinal detachment (Eye disorders) | 1 | 0 | 0 — Not related
Gastritis viral (Infections and infestations) | 0 | 1 | 0 — Not related
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1 | 0 — Not related
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 — Not related
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 — Not related

LIMITATIONS AND CAVEATS:
Study excluded patients who were under the age of 18, had uncontrolled glaucoma, were at risk of developing macular edema (diabetic retinopathy), and women of childbearing potential. Therefore, results may not be generalizable to these populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.